CLINICAL TRIAL: NCT06822985
Title: The Efficacy and Safety of QL1706 As Second-line Treatment in Advanced Hepatocellular Carcinoma Patients Refractory to First-line Therapy: a Single-arm, Phase I Study
Brief Title: QL1706 As Second-line Treatment in Patients with Advanced Hepatocellular Carcinoma
Acronym: QL1706
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wan-Guang Zhang (Other)
Collaborators: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLMA-HCC-IIT-101
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: HCC - Hepatocellular Carcinoma
Keywords: QL1706; Immunotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: QL1706 (Experimental): Drug: QL1706
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — Drug: QL1706 7.5 mg/kg administered as IV infusion on Day 1 of each 21-day cycle

SUMMARY:
This is a phase I trial to assess the safety and preliminary efficacy of QL1706 in Treating Advanced Hepatocellular Carcinoma Patients refractory to prior immunotherapy.

DETAILED DESCRIPTION:
Immune checkpoint inhibitors (ICIs) have produced encouraging results in patients with hepatocellular carcinoma (HCC). Nonetheless, single-agent ICIs are effective in only 15% to 20% of HCC patients. According to the phase 3 LEAP-002 trial, lenvatinib combined with pembrolizumab provides a limited survival advantage over lenvatinib. In China, local treatments combined with tyrosine kinase inhibitors (TKIs) and anti-PD-1 antibodies have been used as the first-line treatment of advanced HCC. However, due to the heterogeneity of cancer, patient responses to monotherapy or combination therapy vary considerably, and only some patients benefit from such therapy. Hence, there is an unmet need to investigate the appropriate treatment for the rapidly expanding group of patients with advanced HCC who had tumor progression on prior anti-PD-1 therapies. QL1706 (PSB205) is a single bifunctional MabPair (a novel technical platform) product consisting of two engineered monoclonal antibodies (anti-PD-1 IgG4 and anti-CTLA-4 IgG1), with a shorter elimination half-life (t1/2) for CTLA-4. The Single-arm, single-center study aims to evaluate the safety and efficacy of QL1706 in treating advanced HCC refractory to prior PD-1 immune checkpoint inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate voluntarily and sign informed consent.
2. 18 years ≤ age ≤ 75 years;
3. Child-Pugh liver function score ≤ 7;
4. ECOG PS 0-1;
5. No serious organic diseases of heart, lung, brain, kidney and other organs;
6. Enhanced MRI examination confirmed advanced hepatocellular carcinoma (CNLC stage II and above, Barcelona stage B and above);
7. Puncture biopsy confirming the pathologic type as hepatocellular carcinoma;
8. Disease progression after receiving first-line therapy(Progressed on/relapsed after at least one prior anti-PD-1 treatment).

Exclusion Criteria:

1. Pregnant and lactating women;
2. Suffering from diseases that affect the absorption, distribution, metabolism or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorders, etc.);
3. A history of gastrointestinal bleeding within the previous 4 weeks or a definite predisposition to gastrointestinal bleeding (e.g., known locally active ulcer lesions, fecal occult blood of ++ or more, or gastroscopy if persistent fecal occult blood of +) that has not been treated in a targeted manner, or any other condition that may have caused gastrointestinal bleeding (e.g., severe fundal/esophageal varices) as determined by the investigator;
4. Active infections, including: HIV (HIV1/2 antibody) positive; active hepatitis B (HBsAg positive and abnormal liver function); active hepatitis C (HCV antibody positive or HCV RNA ≥103 copies/ml and abnormal liver function); active tuberculosis; and other uncontrolled active infections (CTCAE V5.0 >2 level);
5. Other significant clinical and laboratory abnormalities that, in the opinion of the investigator, affect the safety evaluation, e.g., uncontrolled diabetes mellitus, immunodeficiency disorders, chronic kidney disease, grade II or higher peripheral neuropathy (CTCAE V5.0), and abnormal thyroid function;
6. Prior use of anti-CTLA-4 antibody drugs.
7. Inability to follow the study protocol to receive treatment or follow up as scheduled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival(mPFS) | From randomization to the first occurrence of disease progression or death from any cause, whichever occurs earlier, assessed up to 1 year
  measured from the date of first treatment to radiographically documented progression according to mRECIST 1.1 or death from any cause (whichever occurs first). Participants alive and without disease progression or lost to follow-up will be censored at the date of their last radiographic assessment.

SECONDARY OUTCOMES:
overall response rate (ORR) measured by mRECIST criteria | rom the date of first treatment to radiographically documented progression according to mRECIST, assessed up to 2 year
  Complete response (CR): Disappearance of any intra-tumoral arterial enhancement in all target lesions; Partial response (PR): At least a 30% decrease in the sum of diameters of viable (enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Stable disease (SD): Any cases that do not qualify for either partial response or progressive disease; Progressive disease (PD): An increase of at least 20% in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since treatment started.
  ORR=CR+PR.
Overall survival (OS) | from the date of first treatment to the date of death from any cause, assessed up to 2 year
  Overall survival (OS): measured from date of first treatment to the date of death from any cause. Participants alive or lost to follow-up will be censored at the date of their last visit.
Disease control rate (DCR) | from the date of first treatment to radiographically documented response according to mRECIST, assessed up to 2 year
  Percentage of patients that had a CR, PR, or SD ≥ 6 months per mRECIST
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 21 days post-the last treatment
  Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes